CLINICAL TRIAL: NCT06944938
Title: The Role of Probiotics and Dietary Interventions in the Treatment of Periodontitis: A Randomized Controlled Clinical Trial
Brief Title: The Role of Probiotics and Dietary Interventions in the Treatment of Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dicle University (Other)
Responsible Party: Principal Investigator, Feray ÇAĞIRAN YILMAZ, associate professor, Dicle University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dicle University Nutrition
Record Dates: First submitted 2025-04-10; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2019-10

CONDITIONS: Periodontal Diseases
Keywords: Periodontitis; probiotics; diet
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Experimental): traditional periodontitis treatment
  Interventions: Procedure: Non-Surgical Periodontal Treatment
- Probiotic group (Experimental): traditional periodontitis treatment + probiotic support
  Interventions: Procedure: Non-Surgical Periodontal Treatment; Dietary Supplement: Probiotic Supplementation
- Probiotic+diet group (Experimental): traditional periodontitis treatment + probiotic support + diet
  Interventions: Procedure: Non-Surgical Periodontal Treatment; Dietary Supplement: Probiotic Supplementation; Other: Probiotic Supplementation + Personalized Diet

INTERVENTIONS:
Procedure: Non-Surgical Periodontal Treatment — Participants in this arm received standard non-surgical periodontal treatment, including scaling and root planing, without any additional supplementation or dietary modification.
Dietary Supplement: Probiotic Supplementation — Participants in this arm received standard periodontal treatment along with a daily probiotic supplement (1 capsule/day, containing 10⁹ CFU of Lactobacillus rhamnosus and Bifidobacterium animalis subsp. lactis) for six consecutive weeks.
  Arms: Probiotic group; Probiotic+diet group
Other: Probiotic Supplementation + Personalized Diet — Participants in this arm received standard periodontal treatment, the same probiotic protocol as the probiotic group, and a personalized anti-inflammatory diet. The diet was developed by a clinical dietitian and emphasized high-fiber, antioxidant-rich, and prebiotic foods. Consumption of refined carbohydrates, added sugars, and trans fats was restricted.
  Arms: Probiotic+diet group

SUMMARY:
The aim of this study is to evaluate the effects of probiotic supplementation and diet-supported probiotic use on periodontal clinical parameters in individuals with periodontitis. A total of 120 female participants aged between 20-60 years, diagnosed with periodontitis and without systemic diseases, were included in the study. Participants are randomly assigned into three groups: a control group (conventional treatment), a probiotic group (conventional treatment + probiotics), and a diet + probiotic group (conventional treatment + probiotics + personalized diet). Clinical evaluations are performed using measurements of probing depth (PD) and clinical attachment loss (CAL), while dietary intake is assessed using three-day food records. The collected data will be analyzed using SPSS 21.0 software, and a p-value <0.05 will be considered statistically significant.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease that results in the destruction of the supporting tissues of the teeth, potentially leading to tooth loss if left untreated. While conventional periodontal treatment focuses on mechanical removal of plaque and calculus, there is increasing interest in adjunctive therapies that target the host response and the oral microbiome.

Probiotic supplementation has been suggested as a potential supportive approach in periodontal therapy, owing to its ability to modulate the microbial balance and reduce inflammation. Moreover, dietary habits-especially the intake of protein, fiber, sugar, and carbohydrates-may influence periodontal health by affecting systemic and local inflammatory responses.

This randomized controlled clinical trial investigates the effects of probiotic supplementation and a personalized anti-inflammatory diet in individuals with periodontitis. A total of 120 female participants aged 20 to 60 years, without systemic diseases, are included. The participants are randomly assigned into three parallel groups:

Control group: conventional non-surgical periodontal treatment

Probiotic group: conventional treatment + probiotic supplementation

Diet + probiotic group: conventional treatment + probiotic supplementation + personalized diet counseling

The intervention period lasts six weeks. Clinical periodontal parameters, including probing depth (PD) and clinical attachment loss (CAL), are assessed at baseline and at the end of the study. Dietary intake is evaluated through three-day food records collected before and after the intervention.

This study aims to explore the potential of integrating probiotics and diet modifications into a holistic periodontal treatment model. Results will be analyzed following data collection and are not included in this section.

ELIGIBILITY:
Inclusion Criteria:

Female participants aged between 20 and 60 years Clinical diagnosis of periodontitis Presence of at least 20 natural teeth Probing depth between 3 mm and 7 mm (mild to moderate periodontitis) No history of systemic diseases Willingness to participate and provide written informed consent

Exclusion Criteria:

Use of antibiotics or probiotics within the past 6 months Current pregnancy or lactation Smoking Presence of systemic conditions such as diabetes or cardiovascular disease Fewer than 20 natural teeth Inability or unwillingness to comply with study procedures

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Probing Depth (PD) from Baseline to 6 Weeks, measured in millimeters (mm) | Baseline and 6 weeks after intervention
  Probing depth will be measured at six sites per tooth using a UNC-15 periodontal probe. The mean PD per participant will be calculated, and group-level data will be reported as mean ± standard deviation (SD). PD represents the distance from the gingival margin to the base of the periodontal pocket.
Change in Clinical Attachment Loss (CAL) from Baseline to 6 Weeks, measured in millimeters (mm) | Baseline and 6 weeks after intervention
  Clinical attachment loss (CAL) will be assessed at six sites per tooth using a UNC-15 periodontal probe. CAL is defined as the distance from the cemento-enamel junction (CEJ) to the bottom of the pocket. The average CAL per participant will be calculated and presented as mean ± SD at the group level.

SECONDARY OUTCOMES:
Change in Nutrient Intake (Protein, Fiber, Sugar, and Carbohydrate) from Baseline to 6 Weeks | Baseline and week 6
  Three-day food records will be collected at baseline and at week 6. Nutrient intake will be analyzed for protein, fiber, sugar, and carbohydrate using validated dietary analysis software. Data will be reported as mean intake (g/day) and compared across groups.
Correlation Between Nutrient Intake and Periodontal Parameters (PD and CAL) at Week 6 | Week 6
  Pearson correlation analysis will be conducted to examine the relationship between dietary intake (fiber, protein, sugar, carbohydrate) and clinical periodontal outcomes (PD and CAL) at 6 weeks. Results will be reported as correlation coefficients (r) with p-values.

CONTACTS AND LOCATIONS:
Locations (1):
- Private Dental Clinic, Elazığ, Turkey, Elazığ, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will be shared with those who request it.

REFERENCES:
- [Derived] Yilmaz FC, Gorgin NC. The role of probiotics and dietary interventions in the treatment of periodontitis: a pilot randomized controlled clinical trial. BMC Oral Health. 2025 Jul 31;25(1):1287. doi: 10.1186/s12903-025-06510-4. PMID 40745652
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/12345678/